CLINICAL TRIAL: NCT05761249
Title: Observation of Clinical Routine Care for Heart Failure Patients Implanted With BIOTRONIK CRT Devices - HeartInsight Substudy
Brief Title: BIOSTREAM.HF HeartInsight
Status: Completed | Type: Observational
Sponsor: Biotronik SE & Co. KG (Industry)
Responsible Party: Sponsor
Other Study IDs: CR033
Record Dates: First submitted 2023-02-07; First posted 2023-03-09 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-08

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: HeartInsight activation — HeartInsight is activated at enrollment. The attending physicians are free on how to integrate HeartInsight in the patient care. Any treatment is based on routine care according to guidleines. Only documentation occurs on how the physicians use HeartInsight and actions taken in response to HeartInsight alerts

SUMMARY:
The main goal is to learn how HeartInsight is used in clinical routine care. HeartInsight is a heart failure monitoring and notification tool within BIOTRONIK's Home Monitoring System. HeartInsight combines patient data as collected by the implanted devices to alert the attending physicians to impending worsening of heart failure events of the patients. This study will create a sound and seamless documentation of approximately 150 HeartInsight alerts, their processing, subsequent interventions and disease progressions. The data will be analyzed to characterize and quantify the use of HeartInsight in a clinical routine set-up.The patient population consists of heart failure patients with BIOTRONIK CRT-D devices that support HeartInsight.

ELIGIBILITY:
Inclusion Criteria:

* Patient willing and able to give consent
* Participation in BIO|STREAM.HF
* HeartInsight-capable CRT-D device implanted or planned to be implanted
* Symptomatic heart failure NYHA class II or III within 45 days prior to enrollment
* HeartInsight score available or planned use of HeartInsight
* History of worsening of heart failure hospitalization or unscheduled outpatient visit with intravenous diuretic therapy for acute worsening of heart failure
* Patient is willing and able to utilize BIOTRONIK Home Monitoring via CardioMessenger and has sufficient mobile network coverage

Exclusion Criteria:

* Patient with permanent atrial fibrillation or 100% atrial pacing
* Patient is not implanted with an atrial or DX lead or atrial sensing is deactivated
* History of patient incompliance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HeartFailure patients will be recruited by their primary care clinic based on the in/exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2023-05-02 (Actual); Primary Completion 2025-07-09 (Actual); Study Completion 2025-07-09 (Actual)

PRIMARY OUTCOMES:
Rate of WHF hospitalization after HeartInsight activation | through study completion, an average of 1.5 years
  Calculation of worsening heart failure hospitalization events per patient year during study participation when HeartInsight is active

CONTACTS AND LOCATIONS:
Locations (7):
- Czechia (2):
  - Nemocnice Ceske Budejovice, a.s., České Budějovice
  - Fakultní nemocnice Olomouc, Olomouc
- CHU de Brest, Brest, France
- Hungary (2):
  - Semmelweis University, Budapest
  - The University of Pécs, Pécs
- Pauls Stradins Clinical University Hospital, Riga, Latvia
- Hospital de Santa Maria, Lisbon, Portugal

IPD SHARING:
Plan to Share IPD: No